CLINICAL TRIAL: NCT00517907
Title: Phase I Clinical Trial to Assess Safety of Synthetic Preimplantation Factor (PIF-1) in Patients With Steroid-Resistant Acute Graft-Versus-Host Disease (GVHD) After Allogeneic Hematopoietic Stem-Cell Transplantation
Brief Title: Safety Study of Preimplantation Factor (PIF-1) to Treat Acute Steroid-Resistant Graft-Versus-Host Disease (GVHD)
Acronym: PIF1GVHD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: BioIncept LLC (Industry)
Responsible Party: Reuven Or, MD, Bone Marrow Transpl., Cancer Immunother. & Immunobio. Res. Ctr., Hadassah Univ. Hosp.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIF1BMT-HMO-CTIL
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2008-08

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease

ARMS (1):
- 1 (Experimental): 6 steroid-resistant acute GVHD patients, post-matched BMT (serial)
  Interventions: Drug: Preimplantation factor (PIF-1)

INTERVENTIONS:
Drug: Preimplantation factor (PIF-1) — The study will include 6 patients and will last for at least six months. The first three patients will receive PIF-1 (0.5 mg/kg/day for 14 days) by subcutaneous injection. The dosage in the next three patients may be increased to 1 mg/kg/day for 14 days.
  Patients will be treated serially: each patient will be followed for 2 weeks after cessation of PIF-1 administration before the next patient begins PIF-1 administration.

SUMMARY:
The primary goal of this study is to determine the safety and tolerability of a novel peptide - preimplantation factor (PIF-1) - in patients who develop acute steroid-resistant graft-versus-host disease (GVHD) after matched bone marrow transplant (BMT).

Following matched BMT, patients will be placed on standard GVHD preventive therapy (cyclosporine); those who do not respond to cyclosporine are placed on a high-dose steroid regimen for 3 days. Patients that do not respond to this standard treatment will be given PIF-1 subcutaneously for 14 days.

Clinical data and samples will be collected, during PIF-1 administration and for an additional three months thereafter, to examine the long-term effect of PIF-1 treatment on the patients' GVHD status.

DETAILED DESCRIPTION:
Allogeneic BMT is a well-established treatment modality for malignant and non-malignant hematological diseases. Mature donor T cells within the stem-cell graft are the main mediators of the beneficial immune effects, but they are also responsible for the induction of GVHD, which becomes the major cause of morbidity and mortality post-transplant. Acute GVHD occurs within a 100-day period post-transplant and generally is manifested by dermatitis, enteritis, and hepatitis. The treatment of GVHD continues to be a challenge. To eliminate undesirable host-derived hematopoietic elements before BMT, patients are traditionally treated with myeloablative conditioning regimens involving high-dose chemotherapy and total-body irradiation. Standard GVHD prophylaxis and therapy comprise drugs that cause generalized immune suppression and place patients in danger of opportunistic infections and tumor relapse. For acute GVHD prevention, cyclosporine is often used; however, it is frequently necessary to administer long-term high-dose steroids as well.

An acute GVHD patient's lack of response to steroids is associated with poor prognosis. The ideal prophylaxis treatment for BMT patients would be one that prevented the graft from attacking the host, and that modulated the host's immune response so that it would accept the transplant, while maintaining its ability to protect the body against opportunistic hostile agents.

Pregnancy is an immune paradox: it allows maternal (host) acceptance of a semi-allograft (embryo), while it does not cause graft-versus-host or host-versus-graft reactions against the host/mother, or immune suppression. Therefore, the pregnant immunological status is compatible with the desired immune profile in patients undergoing BMT. By replicating the immune profile present in pregnancy in BMT patients, we may be able to reduce the occurrence of GVHD-related morbidity and mortality rates.

Preimplantation factor (PIF-1) is a novel, embryo-secreted peptide whose synthetic version matches the native peptide's properties. PIF-1 appears to play an important role in mediating the maternal response to pregnancy in mammals. In preclinical studies, PIF-1 has been found to be effective in preclinical BMT-GVHD models, without apparent toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Acute steroid-resistant GVHD post matched BMT

Exclusion Criteria:

* Morbidity unrelated to GVHD

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of PIF-1 in steroid-resistant patients who develop acute GVHD, as evidenced by clinical and laboratory indices | within 90 days after first PIF-1 injection

SECONDARY OUTCOMES:
Therapeutic effect of PIF-1 on participants' acute GVHD status, as determined by comparison with the clinical and laboratory indices before intervention | within 90 days after first PIF-1 injection

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Or, MD, Principal Investigator — Bone Marrow Transplantation, Cancer Immunotherapy & Immunobiology Research Center, Hadassah University Hospital, Ein Kerem, Jerusalem, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel